CLINICAL TRIAL: NCT03394547
Title: PUlsed electroMagnetic Field Treatment for Painful Periods: A Randomised Control Trial
Brief Title: Pulsed Electromagnetic Field Treatment for Painful Periods
Acronym: PUMMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Collaborators: BioElectronics Corporation (Industry)
Responsible Party: Principal Investigator, Thomas Justin Clark, Chief Investigator, Birmingham Women's NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BirmimghamWHC
Record Dates: First submitted 2017-11-22; First posted 2018-01-09 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Participants are allocated to 1 of 3 arms: either treatment with an active device, treatment with a placebo device, or no treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomly allocated to a treatment arm through telephone randomisation. If they are allocated to "no treatment" they will be aware of the management, however if allocated to use of a device the participant and care provider will be blinded to weather it is an active device or placebo device. The outcome assessor will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Treatment (Active Comparator): Treatment for 2 menstrual cycles using the pulsed shortwave therapy Allay® device (BioElectronics Corp, Frederick USA)
  Interventions: Device: Allay
- Placebo (Placebo Comparator): Treatment for 2 menstrual cycles using a placebo device which is identical in appearance to the active device but does not emit any pulsed shortwave therapy.
  Interventions: Device: Placebo
- No treatment (No Intervention): No intervention is given and a menstrual diary is completed for 2 cycles.

INTERVENTIONS:
Device: Allay — pulsed shortwave therapy treatment for painful periods
  Arms: Active Treatment
Device: Placebo — A placebo device is given which is identical to the Allay device but emits no pulsed shortwave therapy.
  Arms: Placebo

SUMMARY:
A single-centre, randomised controlled, double blind study comparing use of the Allay pulsed shortwave therapy treatment versus a placebo device or no treatment for management of primary dysmenorrhea.

DETAILED DESCRIPTION:
Women participating in the trial will be randomly allocated to any of the three arms of the study.

* Treatment for 2 menstrual cycles using the PSWT Allay device (BioElectronics Corp, Frederick USA)
* Treatment for 2 menstrual cycles using a placebo device
* No treatment. If they are allocated to a device both the participant and the clinician will be blinded at to weather they are using the active device or the placebo.

Primary Outcome measures are:

* A reduction in dysmenorrhea as measured by the highest pain score on a 10cm visual analogue scale.
* A reduction in average pain score on a 10cm visual analogue scale
* A reduction in use of analgesia as recorded in a pain diary
* Improvement in quality of life as measured through a validated quality of life assessment tool (SF-36 questionnaire)

  - Improvement in menstrual symptoms as recorded through a validated questionnaire (the Modified Menorrhagia Multi-attribute Scale (MMAS)).
* Device acceptability as measured on a 5-point Likert scale ranging from "unacceptable" to "totally acceptable".
* Impact upon associated cyclical symptoms as recorded in a patient symptom diary

ELIGIBILITY:
Inclusion Criteria:

* Female with persistent (>3months) cyclical period pain associated with menstruation (defined as 5 or more on VAS).
* Able to give written, Informed consent
* Able to wear device and keep up-to-date records of use
* Agrees to attend follow up
* If currently using hormonal contraception agrees to continue on the same dose for the duration of the trial.

Exclusion Criteria:

* Age under 16 years.
* Trying to conceive or <6 weeks post partum
* Currently participating or planning to participate in another clinical trial

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
A reduction in dysmenorrhea as measured by the highest pain score on a 10cm visual analogue scale. | 2 months
  Measured as highest pain score on a 10cm visual analogue scale

SECONDARY OUTCOMES:
Impact upon associated cyclical symptoms | 2 months
  Measured through the validated menstrual symptoms questionnaire the Menorrhagia Multi-Attribute Scale
Improvement in quality of life as measured through a validated quality of life assessment tool (SF-36 questionnaire). | 2 months
  Measured through a validated quality of life questionnaire (SF36)
Device acceptability as measured on a 5-point Likert scale ranging from "unacceptable" to "totally acceptable". | 2 months
  Measured by those allocated a device on a 5-point Likert scale ranging from "unacceptable" to "totally acceptable".
Reduction in use of analgesia | 2 months
  Measured through a record of analgesia used during menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Justin Clark, Principal Investigator — Birmingham Women's NHS Foundation Trust
Locations (1):
- University of Birmimgham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided